CLINICAL TRIAL: NCT01803776
Title: The Physical Activity and Nutrition in Children (PANIC) Study
Acronym: PANIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Eastern Finland (Other)
Collaborators: Kuopio University Hospital (Other); University of Jyvaskyla (Other); Kuopio Research Institute of Exercise Medicine (Other); University of Turku (Other); Tampere University (Other); Folkhälsan Researech Center (Other); University of Cambridge (Other); University of Exeter (Other); University of Copenhagen (Other); Norwegian School of Sport Sciences (Other); University of Tromso (Other); University of Iceland (Other); Early Growth Genetics (EGG) Consortium (Unknown); LongITools Consortium (Unknown)
Responsible Party: Principal Investigator, Timo Lakka, Professor of Medical Physiology, University of Eastern Finland
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PANIC
Record Dates: First submitted 2013-02-21; First posted 2013-03-04 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Overweight; Glucose Metabolism Disorders; Lipid Metabolism Disorders; Blood Pressure; Atherosclerosis
Keywords: children; adolescents; physical activity; sedentary time; nutrition; diet; body composition; overweight; obesity; insulin; glucose; lipids; adipokines; myokines; metabolomics; fitness; arterial elasticity; atherosclerosis; blood pressure; bone mineral density; genetics; gene-lifestyle interaction; oral health; oral bacteriomics; wellbeing; depression; sleep; pain; health economics; healthcare services; medication; cost-effectiveness
MeSH Terms: conditions — Overweight; Glucose Metabolism Disorders; Lipid Metabolism Disorders; Atherosclerosis; Motor Activity; Sedentary Behavior; Obesity; Insulin Resistance; Depression; Pain

STUDY DESIGN:
Intervention Model Description: A single-centre controlled trial in which the participants are allocated to a combined physical activity and dietary intervention group and a control group
Oversight: Data Monitoring Committee: No

ARMS (2):
- lifestyle counseling (Experimental): Physical activity and dietary counseling
  Interventions: Behavioral: lifestyle counseling
- Control (No Intervention): No active intervention

INTERVENTIONS:
Behavioral: lifestyle counseling — The physical activity and dietary intervention is based on the Finnish physical activity and dietary recommendations. The children and their parents in the intervention group undergo individualized and family-based physical activity and dietary intervention between the baseline and 2-year follow-up examinations. The children and their parents meet a physical activity specialist and a nutritionist who give detailed and individualized instructions on health promoting physical activity and diet at months 0, 1.5, 3, 6, 12, and 18 with a specific topic at each visit. Between the 2-year follow-up and 8-year follow-up examinations, the intervention continues with yearly physical activity and dietary counseling sessions. The children in the intervention group, particularly those who do not attend organized sports or exercise, will also be encouraged to participate in after-school exercise clubs organized by trained exercise instructors of the study.
  Arms: lifestyle counseling

SUMMARY:
The Physical Activity and Nutrition in Children (PANIC) Study is a single-centre controlled trial on the effects of a combined physical activity and dietary intervention on cardiometabolic risk factors and other health outcomes in a population sample of children from the city of Kuopio, Finland. The study provides novel scientific information for the identification of cardiometabolic diseases and other chronic diseases since fetal period and for the prevention of these chronic diseases since childhood.

The main hypothesis of the PANIC study is that individuals at increased risk of cardiometabolic diseases and other chronic diseases can be identified in childhood and that it is possible to start the prevention of these chronic diseases by a long-term physical activity and dietary intervention since childhood.

DETAILED DESCRIPTION:
We will investigate a population sample of 512 children from the city of Kuopio, Finland. The children will be recruited in 2007-2009 when they are 7-9 years of age and when they will start the first grade in primary schools of the city of Kuopio. The children will be allocated to the combined physical activity and dietary intervention group and the control group after baseline examinations carried out in 2007-2009. The intervention group will undergo individualized and family-based physical activity and dietary intervention, including six intervention visits, for two years. All children from the intervention and control group will be invited to 2-year follow-up examinations carried out in 2009-2011 when they are 9-11 years of age. The intervention group will continue with a less intensive physical activity and dietary intervention until 8-year follow-up examinations carried out in 2015-2017 when the participants are 15-17 years of age. The participants from the intervention and control group will continue with an open follow-up until 14-year follow-up examinations in 2021-2023 when they are 21-23 years of age. All of these study phases will include comprehensive and detailed assessments of behavioral, biological, environmental, and genetic risk factors for cardiometabolic diseases and other chronic diseases. The results of the PANIC Study will help in 1) decreasing the risk of developing cardiometabolic diseases and other chronic diseases since childhood by increasing physical activity, decreasing sedentary time, and improving diet, 2) identifying children and adolescents at increased risk of cardiometabolic diseases and other chronic diseases who would benefit most from the physical activity and dietary interventions, 3) targeting children and adolescents, particularly those at increased risk of cardiometabolic diseases and other chronic diseases, for more careful health examinations, physical activity and dietary interventions, and health follow-up, and 4) preventing cardiometabolic diseases and other chronic diseases as well as their societal consequences in adulthood.

ELIGIBILITY:
Inclusion Criteria:

* boys and girls, 6-9 years of age at baseline, from the city of Kuopio, Finland

Exclusion Criteria:

* physical disabilities that could hamper participation in the intervention
* no time or motivation to attend the study

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 504 (Actual)
Dates: Start 2007-10; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in insulin resistance | From baseline to 2-year follow-up (childhood), 8-year follow-up (adolescence), and 14-year follow-up (early adulthood)
  Fasting serum insulin
Change in fasting plasma glucose | From baseline to 2-year follow-up (childhood), 8-year follow-up (adolescence), and 14-year follow-up (early adulthood)
  Fasting plasma glucose
Change in body composition | From baseline to 2-year follow-up (childhood), 8-year follow-up (adolescence), and 14-year follow-up (early adulthood)
  Body fat percentage and lean body mass assessed by dual-energy X-ray absorptiometry

SECONDARY OUTCOMES:
Change in physical activity | From baseline to 2-year follow-up (childhood), 8-year follow-up (adolescence), and 14-year follow-up (early adulthood)
  Physical activity assessed objectively by heart rate and body movement monitoring
Change in sedentary time | From baseline to 2-year follow-up (childhood), 8-year follow-up (adolescence), and 14-year follow-up (early adulthood)
  Sedentary time assessed objectively by heart rate and body movement monitoring
Change in diet | From baseline to 2-year follow-up (childhood), 8-year follow-up (adolescence), and 14-year follow-up (early adulthood)
  Food consumption and nutrient intake assessed by 4-day dietary recording
Change in cardiorespiratory fitness | From baseline to 2-year follow-up (childhood), 8-year follow-up (adolescence), and 14-year follow-up (early adulthood)
  Maximal workload and peak oxygen consumption assessed by a maximal exercise test on a bicycle ergometer
Change in lipid metabolism | From baseline to 2-year follow-up (childhood), 8-year follow-up (adolescence), and 14-year follow-up (early adulthood)
  Biomarkers of lipid metabolism (fasting triglycerides, HDL cholesterol and LDL cholesterol)
Change in liver adiposity | From baseline to 2-year follow-up (childhood), 8-year follow-up (adolescence), and 14-year follow-up (early adulthood)
  Biomarkers of liver adiposity (alanine aminotransferase and gamma glutamyltransferase)
Change in blood pressure | From baseline to 2-year follow-up (childhood), 8-year follow-up (adolescence), and 14-year follow-up (early adulthood)
  Systolic and diastolic blood pressure at rest
Change in cognitive function | From baseline to 2-year follow-up (childhood), 8-year follow-up (adolescence), and 14-year follow-up (early adulthood)
  General mental ability assessed by Raven's Coloured Progressive Matrices
Change in bone mineral density | From baseline to 2-year follow-up (childhood), 8-year follow-up (adolescence), and 14-year follow-up (early adulthood)
  Change in bone mineral density assessed by dual-energy X-ray absorptiometry
Change in the use of healthcare services | From baseline to 2-year follow-up (childhood), 8-year follow-up (adolescence), and 14-year follow-up (early adulthood)
  Use of healthcare services received from national and local health registries
Change in costs associated with the use of healthcare services | From baseline to 2-year follow-up (childhood), 8-year follow-up (adolescence), and 14-year follow-up (early adulthood)
  Costs associated with the use of healthcare services received from national and local health registries

CONTACTS AND LOCATIONS:
Overall Officials: Timo A Lakka, MD, Principal Investigator — University of Eastern Finland, Kuopio campus
Locations (1):
- University of Eastern Finland, Kuopio, Finland

REFERENCES:
- [Derived] Viisanen M, Raittio E, Ikavalko T, Peltomaki T, Suominen AL, Tolonen V, Soininen S, Karvinen H, Lakka TA. Orthodontic Visits According to Socioeconomic Status Among Children Living in the City of Kuopio, Finland: The PANIC Study. Clin Exp Dent Res. 2026 Feb;12(1):e70280. doi: 10.1002/cre2.70280. PMID 41510745
- [Derived] Liimatta J, Huotari J, du Toit T, Fluck CE, Jaaskelainen J, Hackney AC, Hakkinen MR, Lehtonen M, Auriola S, Lakka TA, Voutilainen R. Serum and hair steroid profiles and their associations with body composition in adolescence. Eur J Endocrinol. 2025 Nov 26;193(6):640-650. doi: 10.1093/ejendo/lvaf235. PMID 41259303
- [Derived] Macro LE, Vlachopoulos D, Haapala EA, Wadey CA, Lakka TA, Barker AR. Effect of Scaling Peak Oxygen Uptake for Body Size and Composition to Assess Cardiometabolic Risk in Children. Med Sci Sports Exerc. 2025 Dec 1;57(12):2795-2806. doi: 10.1249/MSS.0000000000003828. Epub 2025 Jul 25. PMID 40708126
- [Derived] Kraav J, Zagura M, Viitasalo A, Soininen S, Veijalainen A, Kahonen M, Jurimae J, Tillmann V, Haapala E, Lakka T. Associations of Cardiovascular Health Metrics in Childhood and Adolescence With Arterial Health Indicators in Adolescence: The PANIC Study. J Am Heart Assoc. 2024 Nov 19;13(22):e035790. doi: 10.1161/JAHA.124.035790. Epub 2024 Nov 7. PMID 39508145
- [Derived] Aitokari L, Lahti S, Kivela L, Riekki H, Hiltunen P, Vuorela N, Viitasalo A, Soininen S, Huhtala H, Lakka T, Kurppa K. Alanine aminotransferase cutoffs for the pediatric fatty liver disease: Major impact of the reference population. J Pediatr Gastroenterol Nutr. 2024 Mar;78(3):488-496. doi: 10.1002/jpn3.12040. Epub 2023 Dec 10. PMID 38314943
- [Derived] Skinner AM, Barker AR, Moore SA, Soininen S, Haapala EA, Vaisto J, Westgate K, Brage S, Lakka TA, Vlachopoulos D. Cross-sectional and longitudinal associations between the 24-hour movement behaviours, including muscle and bone strengthening activity, with bone and lean mass from childhood to adolescence. BMC Public Health. 2024 Jan 19;24(1):227. doi: 10.1186/s12889-024-17711-x. PMID 38238707
- [Derived] Laamanen SE, Eloranta AM, Haapala EA, Sallinen T, Schwab U, Lakka TA. Associations of diet quality and food consumption with serum biomarkers for lipid and amino acid metabolism in Finnish children: the PANIC study. Eur J Nutr. 2024 Mar;63(2):623-637. doi: 10.1007/s00394-023-03293-8. Epub 2023 Dec 21. PMID 38127151
- [Derived] Liimatta J, Fluck CE, Mantyselka A, Hakkinen MR, Auriola S, Voutilainen R, Jaaskelainen J, Lakka TA. Effects of 2-Year Physical Activity and Dietary Intervention on Adrenarchal and Pubertal Development: The PANIC Study. J Clin Endocrinol Metab. 2023 Nov 17;108(12):e1603-e1613. doi: 10.1210/clinem/dgad367. PMID 37329220
- [Derived] Soininen S, Eloranta AM, Schwab U, Lakka TA. Sources of vitamin D and determinants of serum 25-hydroxyvitamin D in Finnish adolescents. Eur J Nutr. 2023 Mar;62(2):1011-1025. doi: 10.1007/s00394-022-03039-y. Epub 2022 Nov 9. PMID 36350359
- [Derived] Constable AM, Vlachopoulos D, Barker AR, Moore SA, Soininen S, Haapala EA, Vaisto J, Jaaskelainen J, Voutilainen R, Auriola S, Hakkinen MR, Laitinen T, Lakka TA. The Mediating Role of Endocrine Factors in the Positive Relationship Between Fat Mass and Bone Mineral Content in Children Aged 9-11 Years: The Physical Activity and Nutrition in Children Study. Front Endocrinol (Lausanne). 2022 Mar 24;13:850448. doi: 10.3389/fendo.2022.850448. eCollection 2022. PMID 35399927
- [Derived] Kuvaja-Kollner V, Lintu N, Lindi V, Rissanen E, Eloranta AM, Kiiskinen S, Martikainen J, Kankaanpaa E, Valtonen H, Lakka TA. Cost-effectiveness of physical activity intervention in children - results based on the Physical Activity and Nutrition in Children (PANIC) study. Int J Behav Nutr Phys Act. 2021 Sep 6;18(1):116. doi: 10.1186/s12966-021-01181-0. PMID 34488794
- [Derived] Constable AM, Vlachopoulos D, Barker AR, Moore SA, Soininen S, Haapala EA, Vaisto J, Westgate K, Brage S, Mahonen A, Lakka TA. The independent and interactive associations of physical activity intensity and vitamin D status with bone mineral density in prepubertal children: the PANIC Study. Osteoporos Int. 2021 Aug;32(8):1609-1620. doi: 10.1007/s00198-021-05872-z. Epub 2021 Feb 5. PMID 33547487
- [Derived] Lakka TA, Lintu N, Vaisto J, Viitasalo A, Sallinen T, Haapala EA, Tompuri TT, Soininen S, Karjalainen P, Schnurr TM, Mikkonen S, Atalay M, Kilpelainen TO, Laitinen T, Laaksonen DE, Savonen K, Brage S, Schwab U, Jaaskelainen J, Lindi V, Eloranta AM. A 2 year physical activity and dietary intervention attenuates the increase in insulin resistance in a general population of children: the PANIC study. Diabetologia. 2020 Nov;63(11):2270-2281. doi: 10.1007/s00125-020-05250-0. Epub 2020 Aug 20. PMID 32816094
- [Derived] Eloranta AM, Sallinen T, Viitasalo A, Lintu N, Vaisto J, Jalkanen H, Tompuri TT, Soininen S, Haapala EA, Kiiskinen S, Schnurr TM, Kilpelainen TO, Mikkonen S, Savonen K, Atalay M, Brage S, Laaksonen DE, Lindi V, Agren J, Schwab U, Jaaskelainen J, Lakka TA. The effects of a 2-year physical activity and dietary intervention on plasma lipid concentrations in children: the PANIC Study. Eur J Nutr. 2021 Feb;60(1):425-434. doi: 10.1007/s00394-020-02260-x. Epub 2020 May 4. PMID 32367254
- [Derived] Mantyselka A, Lindi V, Viitasalo A, Eloranta AM, Agren J, Vaisanen S, Voutilainen R, Laitinen T, Lakka TA, Jaaskelainen J. Associations of Dehydroepiandrosterone Sulfate With Cardiometabolic Risk Factors in Prepubertal Children. J Clin Endocrinol Metab. 2018 Jul 1;103(7):2592-2600. doi: 10.1210/jc.2018-00184. PMID 29757399
- [Derived] Soininen S, Eloranta AM, Viitasalo A, Dion G, Erkkila A, Sidoroff V, Lindi V, Mahonen A, Lakka TA. Serum 25-Hydroxyvitamin D, Plasma Lipids, and Associated Gene Variants in Prepubertal Children. J Clin Endocrinol Metab. 2018 Jul 1;103(7):2670-2679. doi: 10.1210/jc.2018-00335. PMID 29750416
- [Derived] Mantyselka A, Jaaskelainen J, Eloranta AM, Vaisto J, Voutilainen R, Ong K, Brage S, Lakka TA, Lindi V. Associations of lifestyle factors with serum dehydroepiandrosterone sulphate and insulin-like growth factor-1 concentration in prepubertal children. Clin Endocrinol (Oxf). 2018 Feb;88(2):234-242. doi: 10.1111/cen.13511. Epub 2017 Nov 29. PMID 29112780
- [Derived] Haapala EA, Eloranta AM, Venalainen T, Jalkanen H, Poikkeus AM, Ahonen T, Lindi V, Lakka TA. Diet quality and academic achievement: a prospective study among primary school children. Eur J Nutr. 2017 Oct;56(7):2299-2308. doi: 10.1007/s00394-016-1270-5. Epub 2016 Sep 9. PMID 27612875
- [Derived] Venalainen TM, Viitasalo AM, Schwab US, Eloranta AM, Haapala EA, Jalkanen HP, de Mello VD, Laaksonen DE, Lindi VI, Agren JJ, Lakka TA. Effect of a 2-y dietary and physical activity intervention on plasma fatty acid composition and estimated desaturase and elongase activities in children: the Physical Activity and Nutrition in Children Study. Am J Clin Nutr. 2016 Oct;104(4):964-972. doi: 10.3945/ajcn.116.136580. Epub 2016 Aug 31. PMID 27581473
- [Derived] Collings PJ, Westgate K, Vaisto J, Wijndaele K, Atkin AJ, Haapala EA, Lintu N, Laitinen T, Ekelund U, Brage S, Lakka TA. Cross-Sectional Associations of Objectively-Measured Physical Activity and Sedentary Time with Body Composition and Cardiorespiratory Fitness in Mid-Childhood: The PANIC Study. Sports Med. 2017 Apr;47(4):769-780. doi: 10.1007/s40279-016-0606-x. PMID 27558140
- [Derived] Lintu N, Savonen K, Viitasalo A, Tompuri T, Paananen J, Tarvainen MP, Lakka T. Determinants of Cardiorespiratory Fitness in a Population Sample of Girls and Boys Aged 6 to 8 Years. J Phys Act Health. 2016 Nov;13(11):1149-1155. doi: 10.1123/jpah.2015-0644. Epub 2016 Aug 24. PMID 27334557
- [Derived] Viitasalo A, Eloranta AM, Lintu N, Vaisto J, Venalainen T, Kiiskinen S, Karjalainen P, Peltola J, Lampinen EK, Haapala EA, Paananen J, Schwab U, Lindi V, Lakka TA. The effects of a 2-year individualized and family-based lifestyle intervention on physical activity, sedentary behavior and diet in children. Prev Med. 2016 Jun;87:81-88. doi: 10.1016/j.ypmed.2016.02.027. Epub 2016 Feb 23. PMID 26915641
- [Derived] Haapala EA, Lintu N, Vaisto J, Robinson LE, Viitasalo A, Lindi V, Lakka TA. Associations of Physical Performance and Adiposity with Cognition in Children. Med Sci Sports Exerc. 2015 Oct;47(10):2166-74. doi: 10.1249/MSS.0000000000000652. PMID 26030086
- [Derived] Haapala EA, Poikkeus AM, Kukkonen-Harjula K, Tompuri T, Lintu N, Vaisto J, Leppanen PH, Laaksonen DE, Lindi V, Lakka TA. Associations of physical activity and sedentary behavior with academic skills--a follow-up study among primary school children. PLoS One. 2014 Sep 10;9(9):e107031. doi: 10.1371/journal.pone.0107031. eCollection 2014. PMID 25207813
- [Derived] Vaisto J, Eloranta AM, Viitasalo A, Tompuri T, Lintu N, Karjalainen P, Lampinen EK, Agren J, Laaksonen DE, Lakka HM, Lindi V, Lakka TA. Physical activity and sedentary behaviour in relation to cardiometabolic risk in children: cross-sectional findings from the Physical Activity and Nutrition in Children (PANIC) Study. Int J Behav Nutr Phys Act. 2014 Apr 26;11:55. doi: 10.1186/1479-5868-11-55. PMID 24766669
- See also: Detailed information about the PANIC study from the webpages of University of Eastern Finland — http://www.panicstudy.fi/en/etusivu